CLINICAL TRIAL: NCT02882477
Title: Treatment of Wolfram Syndrome Type 2 With the Chelator Deferiprone, and Incretin Based Therapy
Brief Title: Treatment of Wolfram Syndrome Type 2 With the Chelator Deferiprone and Incretin Based Therapy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, David Zangen, Professor, Hadassah Medical Organization
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0003-16-HMO
Record Dates: First submitted 2016-07-17; First posted 2016-08-29 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes Mellitus; Iron Metabolism Disorders; Gastroduodenal Ulcer; Optic Atrophy; Sensorineural Hearing Loss; Platelet Dysfunction
MeSH Terms: conditions — Diabetes Mellitus; Iron Metabolism Disorders; Peptic Ulcer; Optic Atrophy; Hearing Loss, Sensorineural | interventions — Deferiprone; Acetylcysteine; Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Deferiprone and Acetylcystein (Experimental): PO Deferiprone 20 mg/kg divided in 2 doses PO Acetylcysteine 200 mg divided in 2 doses 5 months duration
  Interventions: Drug: Deferiprone; Drug: Acetylcysteine
- Deferiprone and Acetylcystein with Sitagliptin and Metformin (Experimental): PO Deferiprone 20 mg/kg divided in 2 doses PO Acetylcysteine 200mg divided in 2 doses PO Januet 50/500 if BW < 30kg and 50/850 if BW> 30kg *2/D 5 months duration
  Interventions: Drug: Deferiprone; Drug: Acetylcysteine; Drug: Sitagliptin and Metformin

INTERVENTIONS:
Drug: Deferiprone
  Other Names: Ferriprox
Drug: Acetylcysteine
  Other Names: Reolin
Drug: Sitagliptin and Metformin
  Other Names: Januet
  Arms: Deferiprone and Acetylcystein with Sitagliptin and Metformin

SUMMARY:
Patients who are genetically diagnosed with the recently reported and rare Wolfram syndrome type 2 ( WFS2) and have the degenerative and symptomatic disease including signs such as diabetes, platelet aggregation defect or visual problems will be asked to participate in this study. Knowing the pathomechanism of WFS2 with rapid cell death, after doing baseline investigations to asses the severity of their disease, the participants will be offered a chelator therapy with in addition to the antioxidant Acetylcystein, in diabetic patients an Incertin (GLP-1 ) therapy will be offered as well. The baseline investigations will be repeated after 2 months and after 5 months of therapy in order to asses the progression of the disease and to show if the chelator and anti oxidant therapy and in diabetic patients the GLP-1 therapy could stop the progression of the disease.

DETAILED DESCRIPTION:
In WFS2 mutation the protein nutrient-deprivation autophagy factor-1(NAF-1) is affected.

Given the known result of NAF-1 protein dysfunction in animal and cultured cell line models namely a toxic accumulation of iron in the mitochondria,leading to mitochondrial destruction and oxidative stress we aim to obtain fibroblast samples from the patients and (use laboratory fibroblasts from healthy subjects as controls) These cell cultures will initially be studied for intracellular iron accumulation and then re-evaluated following treatment by Deferiprone and/or Glucagon-like peptide 1 (GLP-1) ex-vivo in the laboratory .

If repeated (n>=3) histological evidence confirms the beneficial effect of Deferiprone and/or GLP-1(incertin based therapy) in the patient's cultured fibroblasts by reversing the toxic iron accumulation in the patient's mitochondria to a normal level, he/she will be offered "in vivo" therapy using the oral chelating agent - with or without dipeptidylpeptidase-4 inhibitor (DPP-4) inhibitors or GLP-1 receptor agonists. Adding GLP-1 based therapy will depend on the diabetic status of the patient.

Prior and following 60 and 150 days of Chelator and/or GLP-1 therapy they will go through the following clinical and laboratory evaluations which will establish the baseline and post therapeutic parameters (outcome) to be compared:

detailed medical history and physical examination complete blood count (CBC) and iron levels platelet aggregation studies Fundoscopy and visual evoked potentials (VEP) Hearing evaluation Oral glucose Tolerance Test optional Intra venous glucose tolerance test (IVGTT) /glucagon/arginine test HBA1C Daily profile of blood glucose Optional CGMS ( continuous glucose monitoring system) Gastroscopy and gastric biopsy if the patient suffers from abdominal pain, hematemesis, melena or iron deficiency anemia or if peptic ulcer disease is clinically suspected.

Based on the routine use of the iron chelator, FDA approved, Deferiprone for Thalassemia (with detailed official guidelines of the Israel association for Pediatric Hematology) and for a similar subcellular iron accumulating disease - e.g. Friedreich Ataxia, we will initially use a dose of 20 mg per kilogram body weight (BW) daily divided in two equal doses. N-Acetylcystein an over the counter drug which also is an anti-oxidant will be given orally in the dose of 200mg twice daily to have a synergistic effect with Deferiprone.

In addition if they suffer from diabetes they will receive Januet (Sitagliptin/metformin) .

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, of any age genetically and clinically diagnosed with Wolfram syndrome type 2.

Exclusion Criteria:

* Patients who are non-cooperative.
* Patients with bone marrow disease or neutropenia.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-05 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Insulin levels in blood in response to Glucose Challenge - Oral Glucose tolerance test (OGTT ) and Intra venous glucose tolerance test (IVGTT) | 5 months
Platelet aggregation to Adenosine diphosphate (ADP) and Collagen - blood test for Platelet function test | 5 months
Nerve conduction velocity in VEP | 5 months
HBA1C level | 5 months
daily glucose level measurement in the blood using Glucometer two to 5 times daily | 5 months
C-Peptide levels in blood in response to Glucose Challenge - Oral Glucose tolerance test ( OGTT ) and Intra venous glucose tolerance test IVGTT | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: David Zangen, Professor, Principal Investigator — Head of pediatric endocrinology department
Locations (1):
- Hadassah medical center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lu S, Kanekura K, Hara T, Mahadevan J, Spears LD, Oslowski CM, Martinez R, Yamazaki-Inoue M, Toyoda M, Neilson A, Blanner P, Brown CM, Semenkovich CF, Marshall BA, Hershey T, Umezawa A, Greer PA, Urano F. A calcium-dependent protease as a potential therapeutic target for Wolfram syndrome. Proc Natl Acad Sci U S A. 2014 Dec 9;111(49):E5292-301. doi: 10.1073/pnas.1421055111. Epub 2014 Nov 24. PMID 25422446
- [Background] Amr S, Heisey C, Zhang M, Xia XJ, Shows KH, Ajlouni K, Pandya A, Satin LS, El-Shanti H, Shiang R. A homozygous mutation in a novel zinc-finger protein, ERIS, is responsible for Wolfram syndrome 2. Am J Hum Genet. 2007 Oct;81(4):673-83. doi: 10.1086/520961. Epub 2007 Aug 20. PMID 17846994
- [Background] Shang L, Hua H, Foo K, Martinez H, Watanabe K, Zimmer M, Kahler DJ, Freeby M, Chung W, LeDuc C, Goland R, Leibel RL, Egli D. beta-cell dysfunction due to increased ER stress in a stem cell model of Wolfram syndrome. Diabetes. 2014 Mar;63(3):923-33. doi: 10.2337/db13-0717. Epub 2013 Nov 13. PMID 24227685
- [Background] Yamane S, Hamamoto Y, Harashima S, Harada N, Hamasaki A, Toyoda K, Fujita K, Joo E, Seino Y, Inagaki N. GLP-1 receptor agonist attenuates endoplasmic reticulum stress-mediated beta-cell damage in Akita mice. J Diabetes Investig. 2011 Apr 7;2(2):104-10. doi: 10.1111/j.2040-1124.2010.00075.x. PMID 24843469
- [Background] Tamir S, Paddock ML, Darash-Yahana-Baram M, Holt SH, Sohn YS, Agranat L, Michaeli D, Stofleth JT, Lipper CH, Morcos F, Cabantchik IZ, Onuchic JN, Jennings PA, Mittler R, Nechushtai R. Structure-function analysis of NEET proteins uncovers their role as key regulators of iron and ROS homeostasis in health and disease. Biochim Biophys Acta. 2015 Jun;1853(6):1294-315. doi: 10.1016/j.bbamcr.2014.10.014. Epub 2014 Oct 23. PMID 25448035
- [Background] Sohn YS, Tamir S, Song L, Michaeli D, Matouk I, Conlan AR, Harir Y, Holt SH, Shulaev V, Paddock ML, Hochberg A, Cabanchick IZ, Onuchic JN, Jennings PA, Nechushtai R, Mittler R. NAF-1 and mitoNEET are central to human breast cancer proliferation by maintaining mitochondrial homeostasis and promoting tumor growth. Proc Natl Acad Sci U S A. 2013 Sep 3;110(36):14676-81. doi: 10.1073/pnas.1313198110. Epub 2013 Aug 19. PMID 23959881
- [Background] Chen YF, Kao CH, Chen YT, Wang CH, Wu CY, Tsai CY, Liu FC, Yang CW, Wei YH, Hsu MT, Tsai SF, Tsai TF. Cisd2 deficiency drives premature aging and causes mitochondria-mediated defects in mice. Genes Dev. 2009 May 15;23(10):1183-94. doi: 10.1101/gad.1779509. PMID 19451219
- [Background] Chen YF, Wu CY, Kirby R, Kao CH, Tsai TF. A role for the CISD2 gene in lifespan control and human disease. Ann N Y Acad Sci. 2010 Jul;1201:58-64. doi: 10.1111/j.1749-6632.2010.05619.x. PMID 20649540
- [Background] Pandolfo M, Hausmann L. Deferiprone for the treatment of Friedreich's ataxia. J Neurochem. 2013 Aug;126 Suppl 1:142-6. doi: 10.1111/jnc.12300. PMID 23859349
- [Background] Drucker DJ. Glucagon-like peptides. Diabetes. 1998 Feb;47(2):159-69. doi: 10.2337/diab.47.2.159. PMID 9519708
- [Background] Yusta B, Baggio LL, Estall JL, Koehler JA, Holland DP, Li H, Pipeleers D, Ling Z, Drucker DJ. GLP-1 receptor activation improves beta cell function and survival following induction of endoplasmic reticulum stress. Cell Metab. 2006 Nov;4(5):391-406. doi: 10.1016/j.cmet.2006.10.001. PMID 17084712
- [Background] Cunha DA, Ladriere L, Ortis F, Igoillo-Esteve M, Gurzov EN, Lupi R, Marchetti P, Eizirik DL, Cnop M. Glucagon-like peptide-1 agonists protect pancreatic beta-cells from lipotoxic endoplasmic reticulum stress through upregulation of BiP and JunB. Diabetes. 2009 Dec;58(12):2851-62. doi: 10.2337/db09-0685. Epub 2009 Aug 31. PMID 19720788